CLINICAL TRIAL: NCT00261274
Title: Evaluation of the Safety of Repeated Autologous Infusions of Enzyme-Converted A-to-O (A-ECO) Red Cells Into Group A Volunteers.
Brief Title: Safety Study of ECO Conversion System For Red Blood Cells.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Velico Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 152-1001
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Anemia
Keywords: transfusion; red blood cells
MeSH Terms: conditions — Anemia | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Group A-ECO (Experimental)
  Interventions: Biological: A-ECO
- Control Group (Placebo Comparator)
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: A-ECO
  Arms: Test Group A-ECO
Biological: Saline
  Arms: Control Group

SUMMARY:
The purpose of this study is to demonstrate that small amounts of a person's own red cells, when treated with an enzyme to make A-ECO Red Blood Cells, can be safely re-infused, repeatedly. Each participant will have some blood drawn, treated with an enzyme, washed and re-infused five times. Additional samples of blood will be drawn for testing and evaluation.

DETAILED DESCRIPTION:
This study will involve a statistically valid number of subjects so that firm conclusions may be drawn about the safety of small volumes of A-ECO cells. All participants will receive their own (autologous) red cells that have been either: 1) treated with an enzyme to create A-ECO cells (test group); or 2) washed with saline (control group). The test and control groups will be compared for the rate and extent any adverse reactions or unexpected laboratory test results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer subjects who have no clinically apparent cardiovascular, renal, pulmonary, endocrinological, autoimmune or neurological disorders
* Blood Group A
* Available for follow up periodically at varying intervals for twelve weeks
* Have a clinical presumption of a stable blood volume
* Between 18 and 65 years of age
* Able to provide informed consent
* Practicing contraception, other than oral or systemically delivered contraceptives, while participating in the study (subjects of potential reproductive age).

Exclusion Criteria:

* Women that are pregnant
* Persons with documented immune deficiencies
* Persons found to have abnormal platelet function or anti-platelet antibodies as determined by a pre-study screen
* Persons with a history of idiopathic thrombocytopenic purpura
* Persons who are bleeding or undergoing an active hemolytic process
* Persons who have any history of hemorrhagic tendency
* Persons who are taking any drug known to interfere with hemostasis, or who take combinations of drugs that have been reported to cause hemostatic problems or interfere with laboratory coagulation and platelet function testing
* Persons who test positive for von Willebrand's disease
* Persons taking investigational drugs or using an investigational device
* Persons with a family history of a bleeding disorder
* Persons with a history of vasculitis
* Persons with a history of a dermatological disorder that might be confused with bruising in the judgement of the investigator
* Persons with medical conditions which represent a contraindication to any study procedure, in the judgement of the investigator
* Persons with unexplained bruising
* Persons with abnormal laboratory screening tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Adverse events, clinically significant bruising over a period of 10 weeks.

SECONDARY OUTCOMES:
Unexpected lab test results over 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Gunter, MD, Study Director — ZymeQuest, Inc.
Locations (6):
- United States (6):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Minnesota, Minneapolis, Minnesota
  - TriCore Reference Laboratories, Albuquerque, New Mexico
  - Hoxworth Blood Center, Cincinnati, Ohio
  - American Red Cross Blood Services-Penn Jersey Region, Philadelphia, Pennsylvania
  - American Red Cross, Norfolk, Virginia

REFERENCES:
- [Background] Goldstein J. Conversion of ABO blood groups. Transfus Med Rev. 1989 Jul;3(3):206-12. doi: 10.1016/s0887-7963(89)70080-8. PMID 2562478
- [Background] Goldstein J, Siviglia G, Hurst R, Lenny L, Reich L. Group B erythrocytes enzymatically converted to group O survive normally in A, B, and O individuals. Science. 1982 Jan 8;215(4529):168-70. doi: 10.1126/science.6274021.
- [Background] Goldstein J. Preparation of transfusable red cells by enzymatic conversion. Prog Clin Biol Res. 1984;165:139-57. No abstract available. PMID 6095313
- [Background] Lenny LL, Hurst R, Zhu A, Goldstein J, Galbraith RA. Multiple-unit and second transfusions of red cells enzymatically converted from group B to group O: report on the end of phase 1 trials. Transfusion. 1995 Nov-Dec;35(11):899-902. doi: 10.1046/j.1537-2995.1995.351196110892.x. PMID 8604485
- [Background] Lenny LL, Hurst R, Goldstein J, Benjamin LJ, Jones RL. Single-unit transfusions of RBC enzymatically converted from group B to group O to A and O normal volunteers. Blood. 1991 Mar 15;77(6):1383-8. PMID 1848117
- [Background] Lenny LL, Goldstein J. The production of group O cells. Biotechnology. 1991;19:75-100. doi: 10.1016/b978-0-7506-9120-8.50009-3. No abstract available. PMID 1664756
- [Background] Lenny LL, Hurst R, Goldstein J, Galbraith RA. Transfusions to group O subjects of 2 units of red cells enzymatically converted from group B to group O. Transfusion. 1994 Mar;34(3):209-14. doi: 10.1046/j.1537-2995.1994.34394196617.x. PMID 8146892
- [Background] Kruskall MS, AuBuchon JP, Anthony KY, Herschel L, Pickard C, Biehl R, Horowitz M, Brambilla DJ, Popovsky MA. Transfusion to blood group A and O patients of group B RBCs that have been enzymatically converted to group O. Transfusion. 2000 Nov;40(11):1290-8. doi: 10.1046/j.1537-2995.2000.40111290.x. PMID 11099655